CLINICAL TRIAL: NCT05790629
Title: Three Dimensional Evaluation of Apexogenesis of Immature Young Permanent Teeth With Different Endodontic Tri-calcium Silicate-Based Putties: Randomized Clinical Trial
Brief Title: Three Dimensional Evaluation of Apexogenesis of Immature Young Permanent Teeth With Different Endodontic Material
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa M Eldehna, lecturer of Pediatric dentistry, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-PD-22-26
Record Dates: First submitted 2023-02-01; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Deep Carious Young 1st Permanent Molar With Open Apex

STUDY DESIGN:
Who Masked: Participant
Masking Description: children do not know which material used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (I) control (Active Comparator): young permanent pulpy exposed carious tooth of the selected participants will be treated with specific technique called apexogenesis using bio-compatible material (endo-sequence putty ). This material is administrated to the tooth by placing about 2-4 mm bulk of material in the pulp champers at the cervical line then sealing the capping material with glass ionomer and stainless steel crown.
  Interventions: Procedure: endo-sequence putty
- Group (II) (Experimental): young permanent pulpy exposed carious tooth of the selected participants will be treated with specific technique called apexogenesis using bio-compatible material (neo-MTA putty). This material is administrated to the tooth by placing about 2-4 mm bulk of material in the pulp champers at the cervical line then sealing the capping material with glass ionomer and stainless steel crown.
  Interventions: Procedure: neo-MTA putty

INTERVENTIONS:
Procedure: endo-sequence putty — pupal medicament which is materials used in case of vital pulp therapy (VPT) procedure after opening access in the inflamed pulp to maintain it is vitality, inducing dentin bridge formation and encourage continued root maturation.
  Other Names: Endodontic Tri-calcium Silicate-Based Puty
  Arms: Group (I) control
Procedure: neo-MTA putty — pupal medicament which is materials used in case of vital pulp therapy (VPT) procedure after opening access in the inflamed pulp to maintain it is vitality, inducing dentin bridge formation and encourage continued root maturation.
  Other Names: Endodontic Tri-calcium Silicate-Based Puty
  Arms: Group (II)

SUMMARY:
Randomized Clinical Trial using Three Dimensional Evaluation of Apexogensis of immature young permanent teeth with Different Endodontic Tri-calcium Silicate-Based Putties

DETAILED DESCRIPTION:
Treatment of immature permanent teeth has always been challenging in endodontics, not only because of their wide-open root apices but also because of the thin underdeveloped dentinal walls.Apexogenesis falls under the category of vital pulp therapy (VPT) procedure to maintain pulp vitality, induce dentin bridge formation and encourage continued root maturation.

To overcome the drawbacks of tricalcium silicate-based cements, a range of bioactive endodontic cements have been developed.

EndoSequence BC RRM-Fast Set Putty and NeoPutty (NuSmile, Houston, TX, USA) are the two materials evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* First permanent molar with pulpitis.
* Sufficient tooth structure for placing rubber dam.
* Presence of open apex.
* Short root length.

Exclusion Criteria:

* Insufficient tooth structure that need post and core.
* Presence of swelling.
* Presence of sinus tract.
* Presence of root fracture.
* Presence of root crack.
* Presence of external or internal root resorption.
* Presence of periapical pathosis.
* Presence of root calcification.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
asymptomatic | one year
  pain relief after procedure by Numeric rating scales on follow up visits.Most pain scales use numbers from 0 to 10. A score of 0 means no pain, and 10 means the worst pain you have ever felt.

SECONDARY OUTCOMES:
complete root maturation | one year
  increasing the length the root till the apex closure which is determined by cone beam analysis

OTHER OUTCOMES:
maintain pulp vitality | one year
  Positive response to sensibility testing. it evaluates the condition of the Pulp Being Very Responsive to a hot and cold Stimulus The pulp is deemed normal when there is a response to the stimulus. Pulpitis is present when there is an exaggerated response that produces pain. The absence of responses to sensibility tests is usually associated with the likelihood of pulp necrosis, the tooth is pulpless,

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university dental clinics and 6 October university dental clinics, Cairo, Choose A State Or Province, Egypt

IPD SHARING:
Plan to Share IPD: No
Three Dimensional Evaluation of Apexogenesis of immature young permanent teeth with Different Endodontic Tri-calcium Silicate-Based Putties: Randomized Clinical Trial